CLINICAL TRIAL: NCT03485014
Title: A Phase 1, Open-Label Study to Evaluate the Pharmacokinetics and Safety of Local Administration of EXPAREL for Postsurgical Analgesia in Pediatric Subjects 12 to Less Than 17 Years of Age
Brief Title: Study in Pediatric Subjects Evaluating Pharmacokinetics and Safety of EXPAREL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-120
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: EXPAREL 4 mg/kg (Experimental): Single dose of EXPAREL 4 mg/kg
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Exparel — EXPAREL 4 mg/kg

SUMMARY:
Primary objective: The primary objective of this study is to evaluate the pharmacokinetics (PK) of EXPAREL in pediatric subjects 12 to less than 17 years of age undergoing spinal surgery.

Secondary objective: The secondary objective of this study is to evaluate the safety of EXPAREL in pediatric subjects 12 to less than 17 years of age undergoing spinal surgery.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, open-label study designed to evaluate the safety and PK profile of EXAPREL when administered intraoperatively at the end of surgery via local infiltration. Fifteen pediatric subjects 12 to less than 17 years of age undergoing spinal surgeries are planned for enrollment.

Subjects will be screened within 30 days prior to study drug administration. During the screening visit, subjects will be assessed for past or present neurologic, cardiac, and general medical conditions that, in the opinion of the investigator, would preclude them from study participation.

Subjects will undergo their pre-planned spinal surgeries per the institution's standard of care. On Day 1, eligible subjects will receive a single dose of EXPAREL 4 mg/kg intraoperatively at the end of surgery via local infiltration into the surgical site. There is no required length of stay in the hospital; subjects may be discharged based on the medical judgment of the treating physician.

A follow-up phone call will be scheduled for all subjects on Day 7. A final follow-up visit will be made on Day 30 to all subjects who received study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects whose parent(s) or guardian(s) has/have signed and dated an informed consent form for the subject to participate in the study, and subjects who have provided written assent to participate in the study (if capable).
2. American Society of Anesthesiologists (ASA) Class 1-3.
3. Male or female subjects 12 to less than 17 years of age on the day of surgery.
4. Body mass index (BMI) at screening within the 20th to 80th percentile for age and sex.
5. A pregnancy test for female subjects of childbearing potential will be conducted in the preoperative holding area according to the study site's standard of care. A negative result for the pregnancy test must be available prior to the start of surgery.
6. Subjects and their parent(s)/guardian(s) must be able to speak, read, and understand the language of the ICF and any instruments used for collecting subject-reported outcomes in order to enable accurate and appropriate responses to study assessments, and provide informed consent/assent.
7. Subjects must be able to adhere to the study visit schedule and complete all study assessments.

Exclusion Criteria:

1. Contraindication to bupivacaine or other amide-type local anesthetics or to opioid medication.
2. Administration of EXPAREL or bupivacaine HCl within 30 days prior to study drug administration.
3. Subjects with coagulopathies or immunodeficiency disorders.
4. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

   In addition, the subject will be ineligible to receive study drug if the following criterion is met during surgery:
5. Any clinically significant event or condition uncovered during the surgery (eg, excessive bleeding, acute sepsis) that might render the subject medically unstable or complicate the subject's postsurgical course.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
AUC of EXPAREL concentration | 0-96 hours
  Area under the concentration curve for EXPAREL

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events and serious adverse events | 0-30 days
  Incidence of treatment-emergent adverse events and serious adverse events through 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Ballock, MD, Principal Investigator — The Cleveland Clinic; Igor Grachev, MD, PhD, Study Director — Pacira Pharmaceuticals, Inc
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States